CLINICAL TRIAL: NCT00912535
Title: Quetiapine Augmentation for Primary Anxiety Disorder or Mood Disorders With Comorbid Anxiety Symptoms
Brief Title: Quetiapine Augmentation for Primary Anxiety Disorder or Mood Disorders With Co-morbid Anxiety Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Chih-Ken Chen, Attending Physician, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1443C00026
Record Dates: First submitted 2009-05-24; First posted 2009-06-03 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Primary Anxiety Disorders; Mood Disorders With Comorbid Anxiety Symptoms
Keywords: Primary Anxiety Disorders; Mood Disorders with Comorbid Anxiety Symptoms

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Quetiapine extended release tablet (Active Comparator): Quetiapine orally at a flexible dose fo 50-300mg/day according to the judgment by the investigator for 8 weeks, as adjunct to the same antidepressant at the same dose.
  Interventions: Drug: Quetiapine extended release tablet
- Placebo (Placebo Comparator): Placebo orally, as adjunct to the same antidepressant at the same dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quetiapine extended release tablet — Quetiapine extended release tablet of 50-300mg/day
  Arms: Quetiapine extended release tablet
Drug: Placebo — Placebo orally, as adjunct to the same antidepressant at the same dose.
  Arms: Placebo

SUMMARY:
The objectives of this study are to evaluate the efficacy and safety of quetiapine extended release tablet versus placebo as adjunct to selective serotonin reuptake inhibitors/serotonin/norepinephrine reuptake inhibitors (SSRI/SNRI) in the augmentation treatment of patient with primary anxiety disorders or mood disorders with co-morbid anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* A diagnosis of primary anxiety disorder or mood disorder with co-morbid anxiety symptoms by Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition (DSM-IV)
* A 14-item Hamilton Anxiety Scale (HAM-A)>= 14
* Subject have received single antidepressant at a therapeutic dose for at least 6 weeks
* Male or female aged 18-65 years
* Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrollment
* Able to understand and comply with the requirements of the study and sign informed consent

Exclusion Criteria:

* Pregnancy or lactation
* Any DSM-IV Axis I disorder not defined in the inclusion criteria.
* Receiving any anti-psychotic 7 days prior to entering the study
* Patients who, in the opinion of the investigator, post an imminent risk of suicide or a danger to self or others
* Known intolerance or lack of response to quetiapine fumarate, as judged by the investigator
* Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrollment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
* Use of any of the following cytochrome P450 3A4 inducers in the 14 days preceding enrollment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St.John's Wort, and glucocorticoids
* Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomization
* Substance or alcohol dependence at enrollment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
* Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrollment
* Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
* Unstable or inadequately treated medical illness (e.g. congestive heart failures, angina pectoris, hypertension) as judged by the investigator
* Involvement in the planning and conduct of the study
* Previous enrollment or randomization of treatment in the present study
* Participation in another drug trial within 4 weeks prior enrollment into this study or longer in accordance with local requirements
* A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:

  * Unstable DM defined as enrollment glycosylated hemoglobin(HbA1c)> 8.5%
  * Admitted to hospital for treatment of DM or DM related illness in past 12 weeks.
  * Not under physician care for DM
  * Physician responsible for patient's DM care has not indicated that patient's DM is controlled
  * Physician responsible for patient's DM care has not approved patient's participation in the study
  * Has not been on the same dose of oral hypoglycaemic drug(S) and/or diet for the 4 weeks prior to randomization. For thiazolidinediones(glitazones) this period should not be less than 8 weeks
  * Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks
* An absolute neutrophil count (ANC) of <= 1.5x10(9) per liter

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Hamilton Anxiety Scale(HAMA-A) total score | 2 months
  From baseline to Week 1, Week 4 and Week 8

SECONDARY OUTCOMES:
Item scores for Abnormal Involuntary Movement Scale(AIMS) | 2 months
  From baseline to Week 1, Week 4 and Week 8
Item scores of Barnes-Akathisia Rating Scale (BARS) | 2 months
  From baseline to Week 1, Week 4 and Week 8
Item scores of Simpson-Angus Scale(SAS) | 2 months
  From baseline to Week 1, Week 4 and Week 8
Body Weight | 2 months
  From baseline to Week 1, Week 4 and Week 8
Vital signs | 2 months
  From baseline to Week 1, Week 4 and Week 8
Adverse event/Serious adverse event | 8-9 weeks
  From the time Informed Consent has been obtained to Week 1, Week 4 and Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Ken Chen, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital - Keelung, Keelung, Taiwan

REFERENCES:
- [Derived] Chen YC, Chen CK, Wang LJ. Quetiapine fumarate augmentation for patients with a primary anxiety disorder or a mood disorder: a pilot study. BMC Psychiatry. 2012 Sep 29;12:162. doi: 10.1186/1471-244X-12-162. PMID 23020711